CLINICAL TRIAL: NCT04456088
Title: Inhaled NO for the Treatment of COVID-19 Caused by SARS-CoV-2
Brief Title: Inhaled NO for the Treatment of COVID-19 Caused by SARS-CoV-2 (CANADA Trial)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated (halted prematurely)
Sponsor: Beyond Air Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAI_COV19_01_CAN
Record Dates: First submitted 2020-07-01; First posted 2020-07-02 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-07

CONDITIONS: COVID-19; SARS-CoV 2; Respiratory Disease; Pneumonia, Viral; Corona Virus Infection
MeSH Terms: conditions — COVID-19; Respiration Disorders; Pneumonia, Viral; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: This is a two phase study. The first 10 subjects will be treated with 80ppm NO; The remaining 40 subjects will be randomized in 1:1 ratio with subjects receiving 150 NO+SST or the SST alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1- Nitric oxide treatment- 80ppm (Experimental)
  Interventions: Combination Product: 80 ppm Nitric Oxide delivered through LungFit Delivery System
- Phase 2- Group 1- Nitric oxide treatment- 150ppm (Experimental)
  Interventions: Combination Product: 150 ppm Nitric Oxide delivered through LungFit Delivery System
- Phase 2- Group 2- control (No Intervention): Standard of Care

INTERVENTIONS:
Combination Product: 150 ppm Nitric Oxide delivered through LungFit Delivery System — Nitric Oxide delivered via LungFit system. Patients will receive inhalations of 150 ppm for 40 minutes 4 time per day plus standard supportive care.
  Arms: Phase 2- Group 1- Nitric oxide treatment- 150ppm
Combination Product: 80 ppm Nitric Oxide delivered through LungFit Delivery System — Nitric Oxide delivered via LungFit system. Patients will receive inhalations of 80 ppm for 40 minutes 4 time per day plus standard supportive care.
  Arms: Phase 1- Nitric oxide treatment- 80ppm

SUMMARY:
The purpose of this open label, 2-phase, study is to obtain information on the safety of 80 ppm and the safety and efficacy of 150 ppm Nitric Oxide given in addition to the standard of care of patients with COVID-19 caused by SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (male and female) admitted to the hospital for COVID-19
2. Patients with oxygen saturation less than 93 % on room air
3. Shortness of breath, with symptom onset within the previous 8 days.
4. Ability to understand and comply with study requirements .
5. Signed informed consent by subject

Exclusion Criteria:

1. Patients who are treated with or require high flow nasal cannula, CPAP, intubation, mechanical ventilation, or tracheostomy
2. Diagnosis of acute respiratory distress syndrome
3. Breastfeeding or pregnancy as evidenced by a positive pregnancy test.
4. Subjects diagnosed with immunodeficiency, with history of congestive or unstable heart disease, left ventricular dysfunction (LVEF <40%) or myocardial damage, severe pulmonary hypertension and/or unstable hypertension
5. History of frequent epistaxis (>1 episode/month).
6. Significant hemoptysis during the last 30 days prior to enrollment
7. Methemoglobin level >3% at screening
8. Patients on systemic steroids (any formulation) within 30 days prior to enrollment.
9. History of daily, continuous oxygen supplementation
10. Patients with BMI greater than or equal to 36
11. Patient receiving drugs that have a contraindication with NO,
12. Patients with clinically significant anemia, e.g., Hb <100 g/L and thrombocytopenia, e.g., Platelets <75 thousand cells/mcL.
13. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data, e.g., known or suspected thalassemia, sickle cell disease or other diseases associated with poor oxygen carrying capacity.
14. The subject is identified by the investigator as being unable or unwilling to perform study procedures.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Time to deterioration | up to 14 days
  Time to deterioration as measured by any one of the following:
  * need for non-invasive ventilation
  * need for high flow nasal cannula (HFNC) or
  * need for intubation
  * Death from any cause

SECONDARY OUTCOMES:
Time to stable oxygen saturation | up to 14 days
  Time to patient having stable oxygen saturation (SpO2) of greater than 92% for longer than 3 hr on room air

OTHER OUTCOMES:
Treatment Emergent Adverse Events and SAEs | 30 days after last inhalation treatment
  Treatment Emergent Adverse Events and SAEs - safety evaluation for 30 days after last inhalation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Asher Tal, MD, Study Director — Beyond Air

IPD SHARING:
Plan to Share IPD: No